CLINICAL TRIAL: NCT02397291
Title: Project 1A) To Determine Whether the Transplacental Gradients for 6 Polyols and Mannose Are Altered in IUGR Pregnancies Compared to Normal Pregnancies. Project 1B) To Determine the Relative Contributions of Transplacental Transport vs. Production by the Conceptus of Both Myoinositol (Major Polyol) and Mannose in IUGR and Normal Pregnancies Using Stable Isotopic Methodology.
Brief Title: Transplacental Gradients and Transport in Intrauterine Growth Restricted (IUGR) Pregnancies Compared to Normal Pregnancies.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 01-517
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: IUGR; Pregnancy
Keywords: Pregnancy; IUGR
MeSH Terms: interventions — Mannose; Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: Measurements of maternal and fetal concentrations (Placebo Comparator): At the time of the elective cesarean section, a blood sample of 0.5 ml will be obtained from a maternal heated hand vein at the time the umbilical cord is clamped. Then, the umbilical cord will be doubly clamped to isolate a segment. The umbilical artery and vein will be sampled for 0.5 ml of blood. There are no stable isotopes infused. Heating the maternal hand vein allows it to be "arterialized." These patients are separate from those required for the stable isotope studies listed below.
  Interventions: Drug: Placebo
- Part 2: Stable Isotope Studies (Active Comparator): Prior to the elective cesarean section, 2 samples from the patient's heated hand vein are obtained to establish a baseline for the compounds. Next, a primed constant infusion containing the stable isotopes of mannose and myoinositol is begun in a peripheral IV of the mother. This is continued approximately 2 hours until the Cesarean section is complete and the umbilical cord samples are obtained. An additional 3 samples are obtained from the patient's heated hand vein: 1 at the start of the cesarean section, 1 at the time the fetus is delivered, and 1 at the time the umbilical cord samples are obtained.
  Interventions: Drug: Mannose; Drug: Myoinositol

INTERVENTIONS:
Drug: Mannose — A primed constant infusion containing the stable isotopes of mannose and myoinositol is administered through a peripheral IV.
  Other Names: D-[U-13C]
  Arms: Part 2: Stable Isotope Studies
Drug: Myoinositol — A primed constant infusion containing the stable isotopes of mannose and myoinositol is administered through a peripheral IV.
  Other Names: D-[U-13C]
  Arms: Part 2: Stable Isotope Studies
Drug: Placebo — placebo
  Arms: Part 1: Measurements of maternal and fetal concentrations

SUMMARY:
The purpose of this study is to determine whether the transplacental gradients for 6 polyols and mannose are altered in intrauterine growth restricted (IUGR) pregnancies compared to normal pregnancies and b) to determine the relative contributions of transplacental transport vs production by the conceptus of both inositol (the major polyol) and mannose in IUGR and normal pregnancies using stable isotopic methodology.

DETAILED DESCRIPTION:
The purposes of this study fall in 2 categories: 1) information important to an understanding of normal pregnancies and the roles of polyols and trace carbohydrates in human fetal nutrition and metabolism and 2) determination of the impact of the small IUGR placenta upon the delivery of polyols and trace carbohydrates to the fetus. Stable isotopes of D-mannose, D-glucose and myoinositol are used to determine the contributions of placental transport of these carbohydrates from the maternal circulation to the fetus vs their synthesis in the fetus and placental tissues. The IUGR pregnancies compare the transport and synthesis of these compounds vs a classification of clinical severity based upon Doppler velocimetry data.

The investigators anticipate that, (just as the investigators have shown for glucose) the fetal enrichment of mannose m+6 will be ~ equal to the maternal enrichment. Thus, without any appreciable dilution of fetal mannose m+6 there is no evidence of fetal production of mannose. This will be further confirmed by the infusion of D-[1-13C]glucose into the maternal circulation. Our previous studies have shown that the fetal enrichment will equal the maternal enrichment. Thus, confirmation will be obtained by comparing the enrichment of fetal mannose m+1 with the fetal enrichment of glucose m+1. The mannose enrichment should be 10% or less of the glucose enrichment. These findings would establish unequivocally that fetal requirements for mannose are met primarily by transplacental transport, not fetal production from glucose.

Conversely, the investigators anticipate demonstrating that the fetal enrichment of myoinositol m+6 is significantly less than the maternal enrichment demonstrating minimal transplacental flux of myoinositol with very little dilution of fetal enrichment by myoinositol production from glucose. This will receive further confirmation by comparing the fetal enrichment of myoinositol m+1 with the fetal enrichment of glucose m+1. For example if the fetal enrichment of myoinositol m+1 is 70% of the fetal enrichment of glucose m+1, then 70% of fetal plasma myoinositol is derived from fetal plasma glucose. This would establish that fetal myoinositol requirements are met by fetal production from glucose rather than by transplacental transport.

ELIGIBILITY:
Inclusion Criteria:

* Normal pregnancy = normal fetal growth by ultrasound, absence of congenital anomalies and no maternal complications.
* IUGR = fetal abdominal circumference < 2 Standard Deviations for gestational age
* Scheduled for elective Cesarean section for clinical indications.
* Age 18-50

Exclusion Criteria:

* Presence of maternal infection, chromosomal abnormalities or congenital anomalies
* Multiple pregnancies
* Emergency Cesarean sections
* Diagnosed with Diabetes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2001-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Galan, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Control Group: At the time of the elective cesarean section, a blood sample of 0.5 ml will be obtained from a maternal heated hand vein at the time the umbilical cord is clamped. Then, the umbilical cord will be doubly clamped to isolate a segment. The umbilical artery and vein will be sampled for 0.5 ml of blood. There are no stable isotopes infused. Heating the maternal hand vein allows it to be "arterialized." These patients are separate from those required for the stable isotope studies listed below.
  Placebo: placebo
- Study Group (IUGR): Prior to the elective cesarean section, 2 samples from the patient's heated hand vein are obtained to establish a baseline for the compounds. Next, a primed constant infusion containing the stable isotopes of mannose and myoinositol is begun in a peripheral IV of the mother. This is continued approximately 2 hours until the Cesarean section is complete and the umbilical cord samples are obtained. An additional 3 samples are obtained from the patient's heated hand vein: 1 at the start of the cesarean section, 1 at the time the fetus is delivered, and 1 at the time the umbilical cord samples are obtained.
  Mannose: A primed constant infusion containing the stable isotopes of mannose and myoinositol is administered through a peripheral IV.
  Myoinositol: A primed constant infusion containing the stable isotopes of mannose and myoinositol is administered through a peripheral IV.
Period: Overall Study
Arm/Group | Placebo/Control Group | Study Group (IUGR)
Started | 19 | 5
Completed | 19 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only Part 1 of this study was started and completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Control Group | Study Group (IUGR) | Total
Number analyzed (Participants) | 19 | 5 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 5 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 5 | 24
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maternal Enrichment of Mannose
Description: The infusion of D-[U-13C]mannose and [U-13C]myoinositol into the maternal circulation is used to establish the degree of transplacental flux of these 2 carbohydrates and to determine if there is evidence of fetal and/or placental production of either of these substrates.
Time Frame: Measured at time of cesarean delivery
Measure: Mean (Standard Deviation); unit: G/DL
Arm/Group | Placebo/Control Group | Study Group (IUGR)
Number analyzed (Participants) | 19 | 5
G/DL | 63.8429 (7.85) | 78.5 (1.97)

2. Primary Outcome: Fetal Enrichment of Mannose
Description: as for outcome 1
Time Frame: Measured at time of cesarean delivery
Measure: Mean (Standard Deviation); unit: G/DL
Arm/Group | Placebo/Control Group | Study Group (IUGR)
Number analyzed (Participants) | 19 | 5
G/DL | 58.54 (20.1) | 76.50 (8.02)

3. Primary Outcome: Maternal Enrichment of Myoinositol
Description: as for outcome 1
Time Frame: Measured at time of cesarean delivery
Measure: Mean (Standard Deviation); unit: G/DL
Arm/Group | Placebo/Control Group | Study Group (IUGR)
Number analyzed (Participants) | 10 | 3
G/DL | 58.543 (19.1) | 76.5 (6.55)

4. Primary Outcome: Fetal Enrichment of Myoinositol
Description: as for outcome 1
Time Frame: Measured at time of cesarean delivery
Measure: Mean (Standard Deviation); unit: G/DL
Arm/Group | Placebo/Control Group | Study Group (IUGR)
Number analyzed (Participants) | 10 | 3
G/DL | 66.8 (17.25) | 59.4 (21.9)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Part 1: Measurements of Maternal and Fetal Concentrations | Part 2: Stable Isotope Studies
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/5
Other Adverse Events (participants affected / at risk) | 0/19 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes